CLINICAL TRIAL: NCT05276583
Title: The Role of Memory Consolidation in Negative Memory Biases in Affective Disorders
Brief Title: Does Depression Impact Our Memory for Rewarding Experiences
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: DMEMxp
Record Dates: First submitted 2021-12-27; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with depression like symptoms: Participants in this condition must indicate that they are currently suffering from a mental health illness and score at least 20 on the Becks Depression Inventory. These participants will undergo the motivate learning task and will study images associated with high and low rewards. After 24-hours participants will be tested on their memory for those images.
  Interventions: Behavioral: Motivated Learning Task
- Healthy controls without depression like symptoms: Participants in this condition must indicate that they do not currently suffer from a mental health condition and score less than 20 on the Becks depression inventory. These participants will also undergo the motivate learning task and will study images associated with high and low rewards. After 24-hours participants will be tested on their memory for those images.
  Interventions: Behavioral: Motivated Learning Task

INTERVENTIONS:
Behavioral: Motivated Learning Task — The Motivated Learning Task is split into two parts, the learning phase, and the test phase. During the learning phase participants are presented with 72 landscape images (targets) which they must memorise. Each image which participants are shown is associated with a reward amount. During the test phase participants are shown the 72 images they saw during the learning phase, known as targets, intermixed with 72 new images they did not see during the learning phase, known as lures. Participants must decide whether the image is "old" (i.e., they saw it during the learning phase) or "new" (i.e. they did not see it during the learning phase). After they have made their old/new decision, participants rate their confidence in their decision on a 3-point scale (i.e., guess, sure, very sure).

SUMMARY:
When individuals experience depression, they may find that their brain does not work in the same way that they are used to. For example, sometimes the ability to remember things that happened during the day is not so good. This might specifically impact positive memories, for example remembering having fun at the ice cream shop with some friends. This is because when individuals are depressed they sometimes can not remember positive experiences as our brains do not have the chemicals needed to store those memories. In this experiment the investigators want to see if the ability to remember positive information is negatively impacted by depression. To do so, participants will look at some images that are related to winning high vs. low rewards. Next they are tested on their memory for those images. Participants will also be asked some questions about themselves and their mental health. The investigators expect that those who are experiencing depression will be less able to remember images related to higher rewards compared to those who are not experiencing depression.

DETAILED DESCRIPTION:
Sleep, at its basis, is known to be an important factor for mental health outcomes, yet the contribution of sleep dependent memory consolidation to those outcomes is poorly understood. In depression, learning and memory consolidation is often impaired and this may have long-term consequences that are driven by poor sleep, for those diagnosed with a depressive disorder. Indeed, depressed patients also have impairments in sleep specific physiological activity, which are crucial for efficient memory consolidation whereby memories are reactivated for long-term storage (e.g., slow-wave-sleep). This may contribute to depression symptoms such as anhedonia, a loss of interest in pleasurable activities, which in one study has been related to reduced ability to remember rewarding experiences and reduced activity in reward-related brain networks (e.g., ventral striatum). In order to understand the complex relationship between, sleep, depression and reward it is first necessary to establish a reliable effect size for the relationship between depression and reward-related memory consolidation. Indeed, in recent years it has been found that many published studies lack statistical power to reliably establish robust effect sizes due to small sample size. Therefore, in this experiment the investigators will examine the impact of depression on reward related memory consolidation with a large sample to yield a reliable estimate of the effect size. All participants will undergo the motivated learning task and will have their memory tested for reward related images before and after a 24-hour retention interval. Based on previous research the investigators predict the following:

H1: Memory for images associated with high reward will be greater compared to memory for images associated with low reward.

H3: Healthy controls will have higher memory performance compared to depressed patients.

H2: The magnitude of the benefit for high reward on memory will be greater for healthy controls compared to depressed patients.

Sample Size:

The investigators determined the sample size by performing a data simulation. They achieved this by simulating effects which are in line with our hypotheses using a linear mixed effects model. That data simulation indicated that 400 participants in total would be required to detect the effects of interest with 95% power. If participants have missing data, then that data will be recollected until the desired sample is achieved.

Procedure

All participants will complete the following procedure online via their choice of browser and computer over two sessions. In the first session participants will first sign the consent form then complete the Becks Depression Inventory (BDI) to determine their mental health status. Once complete participants will provide their demographic information (age, sex, gender, education, etc.), complete the Alcohol Use Disorders Identification Test (AUDIT), the Generalised Anxiety Disorder - 7 (GAD-7), Snaith-Hamilton Pleasure Scale (SHAPS), Stanford Sleepiness Scale (SSS) and lastly the Psychomotor Vigilance Task (PVT). Then participants begin the first part of the Motivated Learning Task, the study phase. After a 24-hour retention interval, participants complete the SSS and PVT a second time then complete the test phase of the Motivated Learning Task. Following the conclusion of the test phase, participants are debriefed.

Analysis Plan:

The investigators will use a linear mixed effects models with maximal effects structures to answer the hypotheses. In this case the maximal structure will be used as not including all slopes, intercepts, and correlation structures can increase false positive rates. However, it is also possible that such a model may not converge due to this. Therefore, if necessary, parameters will be removed iteratively starting with correlations of random slopes and then the random slopes themselves.

To examine the hypotheses (H1, H2 and H3) the following linear mixed effects model will be used and reduced accordingly for the reasons specified above:

d' ~ reward * depression + (reward * depression| participant)

Although there will be a positive effect of reward on memory sensitivity in both depressed participants and healthy controls, the investigators expect that this effect will be more pronounced in the latter.

ELIGIBILITY:
Inclusion criteria

* Prolific approval rating of at least 95% and have participated in at least 10 studies on Prolific.
* Country of residence: United Kingdom
* Aged between 20-45
* Education level: At least A-levels or equivalent
* Participants must use a computer or laptop to participate.
* Participants must not have participated in the study conducted to validate the images used in this experiment and in the experiment from our previous preregistrations.
* Participants must not have participated in the previous studies which used the stimuli for this task.

Exclusion criteria

* Participants who incorrectly answer the practice trials and/or the questions of either the learning or test phases of the Motivated Learning Task. (For every question, they can try twice. Only if they get it wrong twice for a given practice phase/question they are excluded.)
* Participants with reaction times below 150ms in more than 20 % of the flanker task and/or the PVT. (These are considered implausibly fast reaction times that indicate that participants did not participate in the task the way it is intended, e.g., random key presses or clicking)
* who have 20% or more lapses (reaction times above 1000 ms) on the PVT.
* Participants who incorrectly respond on > 50% of the flanker task, indicating they did not pay attention to the task.
* Participants with a d' of 0 and below, indicating chance or worse than chance performance.
* Participants who do not complete both parts of the experiment.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All participants will be recruited online using the online work-sourcing platform Prolific (www.prolific.com). Prolific has access to participant populations who are considered healthy and those who are suffering from mental health conditions. However the website is unable to determine whether participants have depressive symptoms or not, therefore the BDI will be administered to divide participants into healthy controls and those with depressive symptoms as described previously.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Discriminability, d' | immediately after the procedure
  Discriminability refers to the ability of a participant to distinguish between targets, i.e., images that were presented to them, and lures, i.e., images that were not shown to them. This is calculated using the following formula:
  z("hit rate" )-z("false alarm rate")
  and will be calculated for each reward category.

SECONDARY OUTCOMES:
Hit Rate | immediately after the procedure
  The hit rate refers to the number of hits (i.e., correct "old" responses to target images) divided by the number of target trials. The hit rate will be calculated for every reward category.
False Alarm Rate | immediately after the procedure
  The false alarm rate, the number of false alarms (i.e., incorrect "old" responses to lure images)/the number of lure trials. The false alarm rate will be calculated for every reward category
Criterion, C | immediately after the procedure
  Criterion refers to a participants willingness to say "old" irrespective of whether or not they actually saw the image. Criterion is calculate using the following formula:
  (- z("hit rate" )+ z("false alarm rate" )) / 2
  and will be calculated for every reward category.

OTHER OUTCOMES:
Becks Depression Inventory BDI | Assessed at the beginning of the experiment once
  The BDI is a 21-item self-report measure of depression symptoms and will be used to distinguish between groups who are not depressed from those who may suffer from depression. Participants answer with one of four responses per item which is scored from 0 - 3. Scores on the BDI range from 1 - 40 with higher scores being more indicative of severe depression symptoms. Participants who score > 19 will be classified as depressed.
Generalised Anxiety Disorder - 7 GAD | Assessed during the first part of the experiment after the BDI.
  The GAD-7 is a 7-item self-report measure of anxiety, with scores ranging from 0-21, where each item is assigned a score ranging from 0-3. Higher scores are indicative of worse anxiety related symptoms.
Snaith-Hamilton Pleasure Scale (SHAPS) | Assessed during the first part of the experiment after the GAD.
  The SHAPS is a 14-item self-report scale measuring anhedonia. Participants respond with Definitely Agree, Agree, Disagree, and Strongly Disagree to each item, where disagree responses receive a score of 1 and remaining responses receive a score of 0. Scores range from 0 - 14 with higher scores indicating greater levels of anhedonia.
Stanford Sleepiness Scale (SSS) | Assessed during the first and second parts of the experiment, that is before the study phase and before the test phase
  The SSS is a measure of sleepiness that will allow us to rule out whether differences in memory performance between sleep and wake conditions are due to tiredness at learning and test phases. Participants will indicate their sleepiness on a 7-point scale ranging from from 1 = active, vital, alert or wide awake to 7 = no longer fighting sleepiness, about to fall asleep, dream-like thoughts..
Psychomotor Vigilance Task (PVT) | Assessed during the first and second parts of the experiment, that is before the study phase and before the test phase
  Differences in vigilance between healthy and patient conditions will be examined using the 5-minute version of the PVT. Participants are required to press the spacebar whenever they see a timer counting upwards. Vigilance will be assessed by comparing reaction times between session 1 and session 2.
Alcohol Use Disorders Identification Test, AUDIT | The AUDIT is collected during the first part of the experiment before the BDI
  Participants will complete the 10-item self-report version of the AUDIT. In this scale participants indicate their level of alcohol consumption and how often it has impacted their life.

CONTACTS AND LOCATIONS:
Overall Officials: David P Morgan, PhD, Principal Investigator — Central Institute of Mental Health
Locations (1):
- Central Institute of Mental Health, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Once the study has been published all of the anonymised individual participant data will be made available on the Open Science Framework (https://osf.io). The shared data will include all data that underlies the results reported in the publication and supplementary data that may not have been used but may be useful to other researchers. The data will be made available to any researcher who has access to the Open Science Framework and completes a data use agreement form and has IRB or ethical approval to carry out their proposed analyses.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will become available as soon as the findings have been published.
Access Criteria: Researchers will be able to access the data via the Open Science Framework if they have IRB or ethical approval to perform the proposed analyses. Those research must also sign a data use agreement to access the data.

REFERENCES:
- [Background] Adcock RA, Thangavel A, Whitfield-Gabrieli S, Knutson B, Gabrieli JD. Reward-motivated learning: mesolimbic activation precedes memory formation. Neuron. 2006 May 4;50(3):507-17. doi: 10.1016/j.neuron.2006.03.036. PMID 16675403
- [Background] Hoddes E, Zarcone V, Smythe H, Phillips R, Dement WC. Quantification of sleepiness: a new approach. Psychophysiology. 1973 Jul;10(4):431-6. doi: 10.1111/j.1469-8986.1973.tb00801.x. No abstract available. PMID 4719486
- [Background] Roach GD, Dawson D, Lamond N. Can a shorter psychomotor vigilance task be used as a reasonable substitute for the ten-minute psychomotor vigilance task? Chronobiol Int. 2006;23(6):1379-87. doi: 10.1080/07420520601067931. PMID 17190720
- [Background] Snaith P. Anhedonia: a neglected symptom of psychopathology. Psychol Med. 1993 Nov;23(4):957-66. doi: 10.1017/s0033291700026428. PMID 8134519
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Dillon DG, Dobbins IG, Pizzagalli DA. Weak reward source memory in depression reflects blunted activation of VTA/SN and parahippocampus. Soc Cogn Affect Neurosci. 2014 Oct;9(10):1576-83. doi: 10.1093/scan/nst155. Epub 2013 Sep 26. PMID 24078019
- [Background] Button KS, Ioannidis JP, Mokrysz C, Nosek BA, Flint J, Robinson ES, Munafo MR. Power failure: why small sample size undermines the reliability of neuroscience. Nat Rev Neurosci. 2013 May;14(5):365-76. doi: 10.1038/nrn3475. Epub 2013 Apr 10. PMID 23571845
- [Background] Barr DJ, Levy R, Scheepers C, Tily HJ. Random effects structure for confirmatory hypothesis testing: Keep it maximal. J Mem Lang. 2013 Apr;68(3):10.1016/j.jml.2012.11.001. doi: 10.1016/j.jml.2012.11.001. PMID 24403724
- [Background] Bates D, Kliegl R, Vasishth S, Baayen H. Parsimonious mixed models. arXiv preprint arXiv:1506.04967. 2015.
- [Background] Beck AT, Steer RA, Brown GK. Beck depression inventory (BDI-II). Pearson; 1996.
- [Background] Heisig JP, Schaeffer M. Why you should always include a random slope for the lower-level variable involved in a cross-level interaction. European Sociological Review. 2019 ;35(2): 258-79.

DOCUMENTS (1):
  • Informed Consent Form (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/83/NCT05276583/ICF_000.pdf